CLINICAL TRIAL: NCT03948321
Title: Conventional Photodynamic Therapy vs. Painless Photodynamic Therapy for Small Genital Warts：a Randomized, Open-label Trial
Brief Title: Conventional Photodynamic Therapy vs. Painless Photodynamic Therapy for Small Genital Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Dermatology Hospital (Other)
Responsible Party: Principal Investigator, Xiuli Wang, Director, Clinical Professor, Shanghai Dermatology Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-09
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Genital Warts
Keywords: Photodynamic Therapy，PDT; Conventional; Painless; Genital Warts
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluator assesses photographs without prior knowledge of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Painless Photodynamic Therapy（P-PDT） (Experimental): The painless photodynamic therapy（P-PDT）group underwent narrow-band light-emitting diode (LED) irradiation (630 nm; 400 J/cm2) after applying 20% 5-aminolevulinic acid（ALA）cream for 30min. A repeat treatment was administered once weekly for a maximum of 3 weeks.
  Interventions: Procedure: Aminolevulinic acid photodynamic therapy
- Conventional Photodynamic Therapy（C-PDT） (Active Comparator): The conventional photodynamic therapy(C-PDT) group underwent narrow-band light-emitting diode (LED) irradiation (630 nm; 100 J/cm2) after applying 20% 5-aminolevulinic acid cream for 3h.A repeat treatment was administered once weekly for a maximum of 3 weeks.
  Interventions: Procedure: Aminolevulinic acid photodynamic therapy

INTERVENTIONS:
Procedure: Aminolevulinic acid photodynamic therapy — Aminolevulinic acid photodynamic therapy

SUMMARY:
This study is being done to compare a new, continuous illumination and short Incubation time regimen of aminolevulinic acid photodynamic therapy（ALA-PDT) to a conventional regimen for treatment of small genital warts. The hypothesis is that the continuous illumination approach will be less or even no painful, but equally efficacious, as the old regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosed with Genital Warts;
2. Aged > 18 years;
3. All patients are unfit and reluctant to undergo surgery for any reasons, and volunteered to participate in the study and ability to understand and the willingness to sign a written informed consent. Patents agreed to take a picture of the skin lesions.
4. The maximum diameter of a single carcass does not exceed 0.5cm; the skin lesions are at least 6 or more or substantially symmetric

Exclusion Criteria:

1. Those who did not complete the informed consent;
2. The lesions belongs to any of the following conditions: There is damage and inflammation, which may lead to the drug entering the open wound; the individual corpus callosum is more than 0.5cm in diameter; the corpus callosum is located in the vagina, the anal canal, the cervix;
3. Patients with skin photoallergic diseases, porphyria;
4. Known to have a history of allergies to test drugs (porphyrins) and their chemically similar drugs;
5. Patients with other obvious diseases that may affect the evaluation of efficacy; (6)Scars or patients with a tendency to form scars;

(7)Known to have severe immune dysfunction, or long-term use of glucocorticoids and immunosuppressants; (8)Severe heart, liver, kidney disease; with hereditary or acquired People with sexual coagulopathy; (9)Those with severe neurological, psychiatric or endocrine diseases; (10)Women who are pregnant, breast-feeding or using inappropriate contraceptives; those with a history of drug abuse; those who have participated in other drug clinical trials within 4 weeks before treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
The clearance rate of Genital Warts | one week after the last treatment
  The clearance rate of Genital Warts will be measured at one week after the last treatment.

SECONDARY OUTCOMES:
Pain assessment | Immediately, 1st minute, 3rd minute, 5th minute, 7th minute, 10th minute , and every 10 minute to the end of treatment and 2 hours, 12 hours, 24hours and 48 hours after treatment
  The pain will be assessed using Visual Analogue Scale（VAS) with a score range of 0-10. The higher the score, the greater the pain, with 0 being no pain and 10 being the most unbearable pain. Pain will be measured at different time points during and after every treatment ，including immediately, 1st min, 3rd min, 5th min, 7th min, 10th min , and every 10 min to the end of treatment and 2nd h, 12th h, 24th h and 48th h after treatment.
The recurrence rates after treatment | 3 months after the last treatment
  The recurrence rates will be measured at 3 months after the last treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Wang, PhD, MD, Study Chair — Shanghai Skin Disease Hospital
Locations (1):
- Shanghai Dermatology Hospital, Shanghai, Shanghai, Jingan, China, China

IPD SHARING:
Plan to Share IPD: Yes
underlie results
Supporting Information: CSR
Time Frame: One year after finishing this study and for permanency
Access Criteria: anyone who search pubmed